CLINICAL TRIAL: NCT04014959
Title: Mini Theta Burst TMS to Promote Brain Plasticity Indexed by fMRI in MDD Patients
Brief Title: Mini Theta Burst TMS in MDD Patients
Acronym: NARSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Desmond Oathes, Assistant Professor of Psychiatry, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 825761
Record Dates: First submitted 2019-07-01; First posted 2019-07-10 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: depression; TMS; fMRI
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects receive active TMS to their individualized fMRI-guided target. Participants will first receive TMS in the MRI scanner, then over the course of 3-Day TMS Intervention Regimen, and lastly in a final MRI scan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All Participants (Experimental): All participants follow the same procedures.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication. Repetitive TMS (rTMS) is FDA-approved for depression treatment.
  TMS is administered over 5 study visits: an initial TMS/fMRI session, a 3-day TMS intervention regimen, and a post-intervention TMS/fMRI session. During TMS/fMRI sessions, participants receive single pulses of TMS pre/post a short round of Intermittent Theta Burst Stimulation (iTBS), a modified rTMS protocol. Throughout the 3-day intervention regimen, participants receive two full rounds of iTBS daily.
  All study participants receive active TMS.

SUMMARY:
This is not a treatment study.

In this study, the researchers are primarily interested in examining whether functional MRI (fMRI)-guided transcranial magnetic stimulation (TMS) may be more effective than traditional TMS methods at temporarily influencing neural circuit communication. The investigators test this by combining TMS and fMRI technologies to probe and modulate brain activity.

If the novel fMRI-guided TMS stimulation used in this study is more effective than traditional methods, future studies may utilize similar personalized TMS targeting methods to yield even better clinical outcomes.

DETAILED DESCRIPTION:
This study will involve a baseline Magnetic Resonance Imaging (MRI) scan, Transcranial Magnetic Stimulation (TMS), and TMS interleaved with functional MRI (fMRI) scans.

After screening, eligible participants will undergo a 1-hour MRI scan, encompassing structural and functional scans to establish TMS stimulation targets for subsequent visits. During the baseline TMS/fMRI session or pre-intervention TMS/fMRI, single pulses of TMS and a short round of repetitive TMS (rTMS) will be administered to the participant's individualized target while functional MRI scans (fMRI) are collected. Following this, participants will commence a short TMS intervention regimen involving daily rTMS over 3 consecutive days. The day after the intervention, participants will undergo another TMS/fMRI session, or the post-intervention TMS/fMRI, to capture potential changes from the 3-day intervention.

Clinical assessments will be conducted at baseline before the first TMS/fMRI session and again after the final TMS/fMRI session to assess symptom changes.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 60 years old, inclusive
* Right-handed
* Currently experiencing a major depressive episode (MDD)
* Capacity to give informed consent and follow study procedures
* Command of English language to understand/ respond to written and verbal instructions

Exclusion Criteria:

* MRI contraindications (i.e., metal in body, claustrophobia, etc.)
* TMS contraindications (i.e., seizure disorder)
* Diagnosis of exclusionary psychiatric disorder (i.e., schizophrenia, bipolar)
* Current use of psychiatric medication and unable/ willing to safely withdraw
* Refusal to abstain from alcohol or drugs for duration of study
* Medication use that reduces seizure threshold
* Medication that interferes with blood flow (i.e., opioids, antihypertensive)
* Known neurological disorder or significant disability that interferes with study procedures
* Woman who is pregnant or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Oathes, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bossus L, Dickson J, Blaine C, Khalilkhani H, Khan A, Oathes DJ. Causal connectivity maps derived from single-pulse interleaved TMS/fMRI. Sci Rep. 2026 Jan 22;16(1):3070. doi: 10.1038/s41598-025-23684-7. PMID 41571696

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 86 subjects screened for the study, 41 were enrolled and 45 did not start study procedures (32 screen failed, 9 withdrew from participation, and 4 lost to follow-up).
Groups:
- All Participants: All participants follow the same procedures.
  TMS/ fMRI Stimulation: The study uses a modified repetitive TMS stimulation protocol. Participants receive active TMS on five separate days: a baseline TMS/ fMRI scan, three "mini TMS" sessions, and a final TMS/ fMRI scan.
  Again, this level of stimulation is considered to be sub-threshold for that of a TMS treatment protocol.
Period: Baseline MRI and Assessments
Arm/Group | All Participants
Started | 41
Completed | 39
Not Completed | 2
Not completed — Physician Decision | 2
Period: Targeting TMS Scan
Arm/Group | All Participants
Started | 39
Completed | 38
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: TMS + fMRI Scan #1
Arm/Group | All Participants
Started | 38
Completed | 38
Not Completed | 0
Period: Mini TMS Sessions (3 Visits)
Arm/Group | All Participants
Started | 38
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: TMS + fMRI Scan #2
Arm/Group | All Participants
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 41
Age, Continuous [Median (Standard Deviation); unit: years] | 28.9 (9.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Now: Male | 18
  Gender Now: Female | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 23
  More than one race | 4
  Unknown or Not Reported | 2
Snaith-Hamilton Pleasure Scale [Mean (Standard Deviation); unit: units on a scale] — The SHAPS (Snaith et al, 1995) is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Thus, the final score ranges from 0 to 14. Population: Only analyzed participants who completed all study procedures.
  units on a scale
    number analyzed (Participants) | 37
    (all) | 5.84 (3.48)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Evoked Functional Brain Activity Pre/Post Short iTBS Stimulation Before and After the 3-Day TMS Intervention Regimen
Description: Change in subgenual anterior cingulate evoked response (fMRI BOLD) at all four timepoints across the two TMS/fMRI scan sessions: pre-intervention and preceding a single round of iTBS in the scanner (pre-tx, pre-iTBS); pre-intervention, following single iTBS in the scanner (pre-tx, post-iTBS); post intervention, preceding iTBS in the scanner (post-tx, pre-iTBS); and post-intervention, post-iTBS in the scanner (post-tx, post-iTBS).
  Greater negative change is associated with more clinical improvement.
Time Frame: 5 days
Population: Of the 37 participants who completed all study procedures, the data from 36 participants was analyzed. Data one subject was not usable.
Measure: Mean (95% Confidence Interval); unit: % BOLD signal change
Groups:
- All Enrolled Participants: All participants follow the same procedures.
  TMS/ fMRI Stimulation: The study uses a modified repetitive TMS stimulation protocol. Participants receive active TMS on five separate days: a baseline TMS/ fMRI scan, three "mini TMS" sessions, and a final TMS/ fMRI scan.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 36
% BOLD signal change
  Pre-tx/Pre-iTBS | -0.2684097 [-0.3902711 to -0.1465483]
  Pre-tx/Post-iTBS | -0.1897918 [-0.31831449 to -0.06126901]
  Post-tx/Pre-iTBS | -0.2640429 [-0.44510461 to -0.08298111]
  Post-tx/Post-iTBS | -0.4190647 [-0.5876522 to -0.2504772]
Statistical Analysis 1: Comparison: All Enrolled Participants; Statistical analysis of fMRI-guided TMS evoked subgenual anterior cingulate responses (fMRI BOLD) change at Pre-tx/Pre-iTBS. Statistics are from one-sample T-tests vs. 0, 2-tailed. Negative t-values represent negative mean fMRI BOLD percent signal change. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p < 0.001, t-test, 2 sided; t(35)= -4.47
Statistical Analysis 2: Comparison: All Enrolled Participants; Statistical analysis of fMRI-guided TMS evoked subgenual anterior cingulate responses (fMRI BOLD) change at Pre-tx/Post-iTBS. Statistics are from one-sample T-tests vs. 0, 2-tailed. Negative t-values represent negative mean fMRI BOLD percent signal change. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p = 0.005, t-test, 2 sided; t(35)= -3.00
Statistical Analysis 3: Comparison: All Enrolled Participants; Statistical analysis of fMRI-guided TMS evoked subgenual anterior cingulate responses (fMRI BOLD) change at Post-tx/Pre-iTBS. Statistics are from one-sample T-tests vs. 0, 2-tailed. Negative t-values represent negative mean fMRI BOLD percent signal change. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p = 0.005, t-test, 2 sided; t(35)= -2.96
Statistical Analysis 4: Comparison: All Enrolled Participants; Statistical analysis of fMRI-guided TMS evoked subgenual anterior cingulate responses (fMRI BOLD) change at Post-tx/Post-iTBS. Statistics are from one-sample T-tests vs. 0, 2-tailed. Negative t-values represent negative mean fMRI BOLD percent signal change. Alternative hypothesis: true mean is not equal to 0; Test type: Superiority; p < 0.001, t-test, 2 sided; t(35)= -5.05

2. Secondary Outcome: Change in Depression, Anxiety and Stress Scale (DASS-21) Score Pre/Post the 3-Day TMS Intervention Regimen
Description: The Depression, Anxiety, and Stress Scale (DASS-21) is a self-report tool with 21 items, assessing depression, anxiety, and stress levels. The scale scores range from 0 to 63, with higher scores indicating more severe or frequent emotional symptoms. The change in DASS-21 score will be evaluated pre and post the 3-day TMS Intervention Regimen.
Time Frame: Up to one week
Population: Of the 37 participants who completed all study procedures, the data of one subject was unusable. Therefore, the data of 36 participants was used for analysis.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- All Participants: All participants follow the same procedures.
  Transcranial Magnetic Stimulation: Transcranial Magnetic Stimulation (TMS) is a non-invasive form of brain stimulation. TMS can influence activity in various brain regions, and it allows researchers to test or modify brain circuit communication. Repetitive TMS (rTMS) is FDA-approved for depression treatment.
  TMS is administered over 5 study visits: an initial TMS/fMRI session, a 3-day TMS intervention regimen, and a post-intervention TMS/fMRI session. During TMS/fMRI sessions, participants receive single pulses of TMS pre/post a short round of Intermittent Theta Burst Stimulation (iTBS), a modified rTMS protocol. Throughout the 3-day intervention regimen, participants receive two full rounds of iTBS daily.
  All study participants receive active TMS.
Arm/Group | All Participants
Number analyzed (Participants) | 36
score on a scale
  Pre 3-day TMS intervention | 26.78 (1.566064)
  Post 3-day TMS intervention | 17.61 (2.012374)

3. Other Pre Specified Outcome: Change in Evoked Functional Brain Activity Before and After the 3-Day TMS Intervention Regimen
Description: Change in subgenual anterior cingulate evoked response (fMRI BOLD) Before and After the 3-Day TMS Intervention Regimen
  Greater negative change is associated with more clinical improvement.
Time Frame: Up to one week
Population: as for outcome 2
Measure: Mean (Standard Error); unit: % BOLD signal change
Arm/Group | All Participants
Number analyzed (Participants) | 36
% BOLD signal change
  Pre 3-day TMS intervention | -0.19 (0.063308)
  Post 3-day TMS intervention | -0.42 (0.083043)
Statistical Analysis 1: Comparison: All Participants; Analysis to investigate the correlation between changes in DASS-21 Scores (Secondary Outcome) and Evoked Functional Brain Activity (Other Pre-specified Outcome) pre and post the 3-Day TMS Intervention Regimen; Test type: Other — Statistics are an unadjusted linear regression of change in DASS-21 depression score on the pre-intervention TMS/fMRI evoked brain response; p = 0.007, Regression, Linear; β = -33.60

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from study enrollment until study completion (Up to 3 weeks).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 5/41
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=41)
Vomiting during TMS/fMRI scan (Gastrointestinal disorders) | 1 (1) — Participant threw up during TMS/ fMRI scan and said it was due to not eaten all day; after they ate crackers they insisted on finishing rest of scan and had no further issues. Though rare, nausea is listed as a possible side effect of TMS.
Anxiety during TMS/fMRI scan (Psychiatric disorders) | 1 (1) — Subject reported anxiety during TMS/ fMRI scan. Participant took a 15min break and then decided to finish scan.
Emotional Discomfort during assessment (Social circumstances) | 1 (1) — Patient complained of emotional discomfort following the Columbia-Suicide Severity Rating Scale (C-SSRS).
Faint (General disorders) | 1 (1) — Subject had a brief feeling of 'blacking out' and faint feeling during TMS stimulation. Subject was withdrawn from the study for safety.
Cutis verticis gyrata (CVG) (Musculoskeletal and connective tissue disorders) | 1 (1) — After completing the structural scan (T1) staff noticed that subject had unsual folds in their scalp. They were referred to a radiologist who determined they had CVG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04014959/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/59/NCT04014959/ICF_001.pdf